CLINICAL TRIAL: NCT00945269
Title: Phase I/II Study To Evaluate The Safety Of Cellular Adoptive Immunotherapy Using Autologous CD8+ Antigen-Specific T Cell Clones Following CD25 Lymphodepletion For Patients With Metastatic Melanoma
Brief Title: Therapeutic Autologous Lymphocytes, Aldesleukin, and Denileukin Diftitox in Treating Patients With Stage III-IV Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: ONTAK has been pulled off the market for further testing. Subsequently, EISAI will no longer be supporting clinical trials that utilize this drug.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sylvia Lee, Research Associate, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2271.00; NCI-2010-00738 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); K12CA076930 (NIH); R21CA137647 (NIH)
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Recurrent Melanoma; Stage III Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interleukin-2; denileukin diftitox; Biopsy; Immunohistochemistry; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cellular adoptive immunotherapy) (Experimental): Patients receive autologous T-cell IV over 30-60 minutes on days 0 and 28 and low-dose aldesleukin SC twice daily on days 0 to 13 and 28 to 41. Beginning 4-6 days before second T-cell infusion, patients receive denileukin diftitox IV over 30 minutes on days 1-3.
  Interventions: Biological: therapeutic autologous lymphocytes; Biological: aldesleukin; Biological: denileukin diftitox; Procedure: biopsy; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Genetic: polymerase chain reaction

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes — Given IV
  Other Names: AL; Autologous Lymphocytes; autologous T cells
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Biological: denileukin diftitox — Given IV
  Other Names: DAB389 interleukin-2; DAB389 interleukin-2 immunotoxin; DAB389-IL2; DABIL2
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: laboratory biomarker analysis — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR

SUMMARY:
RATIONALE: White blood cells that have been treated in a laboratory may be able to kill tumor cells in patients with melanoma. Aldesleukin and denileukin diftitox may stimulate the white blood cells to kill melanoma cells. Giving therapeutic autologous lymphocyte therapy together with aldesleukin and denileukin diftitox may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects of giving therapeutic autologous lymphocytes together with aldesleukin and denileukin diftitox and to see how well it works in treating patients with stage III-IV melanoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety of cellular adoptive immunotherapy in melanoma patients using autologous CD8+ antigen-specific T-cell clones following CD25 lymphodepletion.

II. Determine the influence of CD25 lymphodepletion on the duration of in vivo persistence of adoptively transferred CD8+ antigen-specific cytotoxic T-cell (CTL) clones.

SECONDARY OBJECTIVES:

I. Assess the anti-tumor efficacy of cellular adoptive immunotherapy in melanoma patients using autologous CD8+ antigen-specific T cell clones following CD25 lymphodepletion.

II. Evaluate the induction of T cells to non-targeted tumor-associated antigens (antigen-spreading) following adoptive transfer of CD8+ antigen-specific CTL and CD25 lymphodepletion.

OUTLINE: This is a phase I study followed by a phase II study.

Patients receive autologous T-cell intravenously (IV) over 30-60 minutes on days 0 and 28 and low-dose aldesleukin subcutaneously (SC) twice daily on days 0 to 13 and 28 to 41. Beginning 4-6 days before second T- cell infusion, patients receive denileukin diftitox IV over 30 minutes on days 1-3. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks, 8 weeks, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological documentation of melanoma
* Expression of human leukocyte antigen (HLA)-A2 or B44 as determined by HLA typing lab
* Patients whose tumor expresses targeted antigen and restricting allele against which CD8 T cell clones can be generated
* Karnofsky Performance status of at least 80% and an expected survival of greater than 6 months
* Bi-dimensionally measurable disease by palpation on clinical exam, or radiographic imaging (X-ray, computed tomography [CT] scan)
* Normal cardiac stress test (treadmill, echocardiogram, or myocardial perfusion scan) within 182 days prior to enrollment is required of patients with a history of cardiac disease
* Pulse > 45 or < 120
* Weight >= 45 kg
* Temperature =< 38C (< 100.4 F)
* White blood cells (WBC) >= 3,000
* Hematocrit (HCT) >= 30%
* Platelets >= 100,000
* Patients must be willing and able to discontinue the use of all antihypertensive medications 24 hours prior to and during IL2 therapy

Exclusion Criteria:

* Pregnant women, nursing mothers, or women of reproductive ability who are unwilling to use effective contraception or abstinence
* Serum creatinine > 1.6mg/dL
* Creatinine clearance < 75 ml/min
* Aspartate aminotransferase (AST) > 2.5 x upper limit of normal
* Alanine aminotransferase (ALT) > 2.5 x upper limit of normal
* Bilirubin > 1.6 or international normalized ratio (INR) > 1.5 due to hepatic dysfunction
* Albumin < 3.0g/dL
* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam; patients so identified will undergo pulmonary functions testing and those with Forced expiratory volume in one second (FEV1) < 80% predicted or diffusing capacity of the lung for carbon monoxide (DLco) (corr for hemoglobin [Hgb]) < 75% will be excluded
* Significant cardiovascular abnormalities as defined by any one of the following: congestive heart failure, symptoms of coronary artery disease
* Symptomatic central nervous system (CNS) metastases greater than 1 cm at time of therapy; patients with 1-2 asymptomatic, less than 1cm brain/CNS metastases without significant edema may be considered for treatment
* Patients with active infections or oral temperature > 38.2 C within 48 hours of study entry or systemic infection requiring chronic maintenance or suppressive therapy
* Chemotherapeutic agents (standard or experimental), radiation therapy, or other immunosuppressive therapies less than 3 weeks prior to T cell therapy)
* Concurrent treatment with steroids
* Patients must not be receiving any other experimental drugs within 3 weeks of the initiation of the protocol and must have recovered from all side effects of such therapy
* The following agents are not allowed while on study: systemic corticosteroids (except as outlined for management of toxicity of nontransduced CTL), immunotherapy (for example, interleukins, interferons, melanoma vaccines, intravenous immunoglobulin, expanded polyclonal TIL or LAK therapy), pentoxifylline, or other investigational agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
In vivo survival of CD8+ transferred T-clones | Days +0, 1, 3, 7, 14, 22, 28, 29, 31, 35, 42, 49, 56, 63, 70, 77, 84
  The design of this trial using the first infusion of CD8 T cells administered alone as a baseline for each patient permits intra-patient analysis using paired samples with increased statistical power.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Lee, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States